CLINICAL TRIAL: NCT07376564
Title: Exploring the Power of Theacrine: Assessing the Impact of High Theacrine Doses on Hemodynamic Measures, Cognitive Measures, and Physiological Stress
Brief Title: Assessing the Impact of High Theacrine Doses on Hemodynamic Measures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Titch Madzima (Other)
Responsible Party: Sponsor-Investigator, Titch Madzima, Associate Professor, Elon University
Organization: Elon University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2791
Record Dates: First submitted 2026-01-18; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hemodynamic Measure; Cognitive Performance in Healthy Volunteers
Keywords: Theacrine; Hemodynamic measures; Cognitive Performance; Cortisol
MeSH Terms: interventions — maltodextrin; 1,3,7,9-tetramethyluric acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): 6 mg/kg Maltodextrin Placebo
  Interventions: Dietary Supplement: Maltodextrin (Placebo)
- Low dose (Experimental): 3mg/kg Theacrine
  Interventions: Dietary Supplement: Low dose theacrine
- Medium dose (Experimental): 6mg/kg Theacrine
  Interventions: Dietary Supplement: Medium dose theacrine
- High dose (Experimental): 9mg/kg Theacrine
  Interventions: Dietary Supplement: High dose theacrine

INTERVENTIONS:
Dietary Supplement: Maltodextrin (Placebo) — 6 mg/kg Maltodextrin Placebo
  Arms: Placebo
Dietary Supplement: Low dose theacrine — 3mg/kg theacrine
  Arms: Low dose
Dietary Supplement: Medium dose theacrine — 6mg/kg theacrine
  Arms: Medium dose
Dietary Supplement: High dose theacrine — 9mg/kg theacrine
  Arms: High dose

SUMMARY:
This project measured physiological and cognitive variables to determine the effectiveness of Theacrine (TCR) as a stimulant at doses greater than those previously tested. The study will be the first TCR study to use doses relative to body weight and will investigate impacts on regular caffeine consumers. A secondary aim of the study is to determine the impact of acute TCR supplementation on salivary cortisol and sAA, two physiological measures of stress and sympathetic nervous system activation. The findings of the study will provide new insight into the effects of higher TCR dosages, contributing to the analysis of TCR as a caffeine alternative for individuals with hypertension, tachycardia, or healthy caffeine consumers wanting to avoid a stimulant with adverse or habitual effects

ELIGIBILITY:
Inclusion Criteria:

- habitual caffeine consumer (≥2 days/week)

Exclusion Criteria:

* existing heart disease or conditions (cardiovascular and/or heart disease, stroke, diabetes hypertension, tachycardia)
* a smoker
* allergy to caffeine or Theacrine
* caffeine sensitivity (negative symptoms such as jitters after consuming low doses)
* pregnant
* on heart or blood pressure medication

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Change in systolic blood and diastolic blood pressure post consumption of theacrine | Pre-consumption, then 60, 90, 120, 150, 180 minutes post-consumption of theacrine
  mmHg change in blood pressure measures
Change in heart rate post consumption of theacrine | Pre-consumption, then 60, 90, 120, 150, 180 minutes post-consumption of theacrine
  beats per minute change in heart rate measure
Changes in executive function as a measure of cognitive performance using the Trail Making Test | Pre-consumption, then 60, 90, 120, 150, 180 minutes post-consumption of theacrine
  Time to completion of the Trail Making Test as a measure of executive function
Changes in attention as a measure of cognitive performance using the Flanker Inhibitory Control and Attention task | Pre-consumption, then 60, 90, 120, 150, 180 minutes post-consumption of theacrine
  Accuracy of congruent and incongruent trials as measures of attention
Changes in focus as a measure of cognitive performance using the Flanker Inhibitory Control and Attention task | Pre-consumption, then 60, 90, 120, 150, 180 minutes post-consumption of theacrine
  Reaction time were recorded as measures of focus

SECONDARY OUTCOMES:
Change in salivary cortisol and alpha-amylase post consumption of theacrine | Pre-consumption, then 60, 90, 120, 150, 180 minutes post-consumption of theacrine
  µg/dL change in cortisol and alpha-amylase levels from baseline as non-invasive measures of physiological stress

CONTACTS AND LOCATIONS:
Overall Officials: Takudzwa A Madzima, PhD, Principal Investigator — Elon University
Locations (1):
- Department of Exercise Science, Koury Athletics Center at Elon University, Elon, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
all individual deidentified participant data that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD data sharing will be available starting 6 months after publication
Access Criteria: The data generated and analyzed during this study will be available starting 6 months after publication upon request from the principal investigator